CLINICAL TRIAL: NCT03608696
Title: Modeled Dose Exposure of Sublingual Buprenorphine in the Neonatal Opioid Abstinence Syndrome
Brief Title: Buprenorphine Pharmacometric Open Label Research Study of Drug Exposure
Acronym: B-PHORE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18C.272
Record Dates: First submitted 2018-06-25; First posted 2018-08-01 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Neonatal Abstinence Syndrome; Neonatal Opiate Withdrawal Syndrome
Keywords: buprenorphine; pharmacometrics
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- buprenorphine (Experimental): Buprenorphine 0.075 mg ml sublingual solution
  Initial daily dose 24 mcg/kg/day Initial unit dose 8 mcg/kg q8 hours Maximum daily dose 75 mcg/kg/day Maximum unit dose 25 mcg/kg q8 hours Up-titration rate 33% Maximum # of up-titrations 4 Weaning rate 15% Cessation (bottom) dose < Initial dose Dosing interval until bottom dose (hrs) 8 Dose interval extension #1 at bottom dose (hrs) 12 Dose interval extension #2 at bottom dose (hrs) 24
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — buprenorphine 0.075 mg/ml solution

SUMMARY:
Neonatal withdrawal syndrome is a series of signs and symptoms in infants exposed to opioids in utero. Buprenorphine has demonstrated a 40% reduction in length of pharmacologic treatment compared to oral morphine. These results were with an empirically derived dose. This study will use pharmacokinetic modeling-informed dosing to clarify the dose/response relationship and use a rational approach to define an optimal dose regimen. The clinical trial will be open label, single arm design with a goal of initial testing of a new dosing regimen.

DETAILED DESCRIPTION:
The overall rationale for this study is to explore new dose regimens in a small number of patients. There is evidence from pharmacometric models with dose simulation that suggest there is room for improvement in buprenorphine dosing. This study will explore these doses. While the endpoint will be primarily pharmacokinetic, it is likely that the revised dose regimen will be more effective and thus holds the potential for benefit for those infants participating. This information will be used to feed back to the model and generate rationally derived, optimal doses to be tested in subsequent efficacy trials.

The neonatal abstinence syndrome (NAS) is a set of signs of withdrawal in an infant with in utero exposure to opioids. Cardinal manifestations include increased muscle tone, autonomic instability, irritability, poor sucking reflex, gastrointestinal symptoms, and impaired weight gain. All infants are treated with non-pharmacologic methods such as swaddling, rooming in with mother and minimization of stimuli. Despite these measures, ~50% of infants require pharmacologic treatment to ensure proper growth and development. While the optimal pharmacologic treatment for NAS has not been identified, expert review identifies an opioid as the primary therapy. In the US 80% of infants are treated with morphine and 20% with methadone. Sublingual buprenorphine has been demonstrated to be safe and effective in an open label phase 1 clinical trial conducted by the Thomas Jefferson University Team [NCT00521248]. These data were used to plan the BBORN (Blinded Buprenorphine OR Neonatal morphine solution) clinical trial [NCT01452789] comparing buprenorphine to morphine for NAS. BBORN demonstrated a 40% reduction in length of treatment compared to morphine in a double blind fashion (New England Journal of Medicine, June 2017). The external validity of this finding has been supported by retrospective examination of buprenorphine used in a treatment paradigm at the University of Cincinnati Medical Center, with a reduction in length of treatment of ~30% in >200 infants.

Dose selection for both the phase 1 trial and the efficacy trial (BBORN) were empirically derived. A population pharmacokinetic model for buprenorphine in NAS has been published by our group. In addition a pre-specified endpoint for the BBORN trial was a pharmacokinetic analysis of buprenorphine. A pharmacokinetic/pharmacodynamic model from the BBORN study has been published (Clinical Pharmacology and Therapeutics, March 2018). The time to control of symptoms was directly tied to buprenorphine exposure, which itself appeared to be driven primarily by clearance. Among the strengths of pharmacometric models is the ability to simulate in silico many potential dose regimens. In this manner, a dose regimen can be chosen that is more likely to be in the desired range of concentrations. This approach also allows for incorporation of covariates of drug exposure or response to treatment. This is much safer and efficient than the traditional approach of choosing an empiric dose that would need to be tested in clinical trial. An ideal dose would quickly reach this exposure while maintaining a good safety margin. There was no evidence of decline in respiratory rate in infants treated with higher doses of buprenorphine compared to lower doses, or those treated with buprenorphine compared to those treated with morphine. This may allow a higher initial dose to more quickly reach therapeutic buprenorphine concentrations. This ultimately could lead to shorter lengths of treatment and stay, though achieving this goal is outside of the scope of the current proposed project.

In summary, buprenorphine at the dose and schedule used in prior clinical trials has been demonstrated to be safe and effective. The goal of the proposed study is to simulate a dose of sublingual buprenorphine for NAS using pharmacometric modelling techniques. This dose will be tested in infants requiring treatment for NAS. Pharmacokinetic samples would be collected and used to confirm and refine the pharmacokinetic model. The proposed study would allow broad examination and refinement of the exposure/response relationship. This optimized dose could later be used in an efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 36 weeks gestation
2. Exposure to opioids in utero
3. Demonstration of signs and symptoms of neonatal abstinence syndrome requiring pharmacologic treatment

Exclusion Criteria:

1. Major congenital malformations and/or intrauterine growth retardation, defined as birth weight <2000 gm
2. Medical illness requiring intensification of medical therapy. This includes but is not limited to suspected sepsis requiring antibiotic therapy.
3. Hypoglycemia requiring treatment with intravenous dextrose
4. Bilirubin >20 mg/dL (The need for phototherapy is not exclusionary)
5. Inability of mother to give informed consent due to co-morbid psychiatric diagnosis

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hosptial, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The sharing plan has not yet been defined
Supporting Information: Study Protocol, SAP, ICF
Time Frame: until 2024
Access Criteria: Consent of principal investigator or designee, with data use agreement in place

REFERENCES:
- [Result] Eudy-Byrne R, Zane N, Adeniyi-Jones SC, Gastonguay MR, Ruiz-Garcia A, Kaushal G, Kraft WK. Pharmacometric dose optimization of buprenorphine in neonatal opioid withdrawal syndrome. Clin Transl Sci. 2021 Nov;14(6):2171-2183. doi: 10.1111/cts.13074. Epub 2021 Sep 16. PMID 34080312

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine: Buprenorphine 0.075 mg ml sublingual solution
  Initial daily dose 24 mcg/kg/day Initial unit dose 8 mcg/kg q8 hours Maximum daily dose 75 mcg/kg/day Maximum unit dose 25 mcg/kg q8 hours Up-titration rate 33% Maximum # of up-titrations 4 Weaning rate 15% Cessation (bottom) dose < Initial dose Dosing interval until bottom dose (hrs) 8 Dose interval extension #1 at bottom dose (hrs) 12 Dose interval extension #2 at bottom dose (hrs) 24
  Buprenorphine: buprenorphine 0.075 mg/ml solution
Period: Overall Study
Arm/Group | Buprenorphine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled subjects are those who required pharmacologic therapy for neonatal opioid withdrawal syndrome
Arm/Group | Buprenorphine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 25.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Pharmacokinetics
Description: Goal is to define buprenorphine pharmacokinetic exposure (Area under the plasma concentration versus time curve (AUC)) in infants treated with buprenorphine for neonatal abstinence syndrome (NAS) using a model-based optimized dose.
Time Frame: Duration of pharmacologic treatment for neonatal abstinence syndrome up to 70 days of age
Population: N/A (PK data was not usable as analyzed for this study as most was below the limit of quantification.)
Arm/Group | Buprenorphine
Number analyzed (Participants) | 0

2. Other Pre Specified Outcome: Number of Participants With Treatment Related Adverse Events
Description: The number of participants with treatment related adverse events
Time Frame: Duration of pharmacologic treatment for neonatal abstinence syndrome, up to 70 days of age
Population: Adverse events in study population
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine
Number analyzed (Participants) | 10
Participants | 2

3. Other Pre Specified Outcome: Length of Treatment
Description: Length of treatment with buprenrophine for NAS (hours) of a model-based optimized dose of buprenorphine for infants treated for NAS.
Time Frame: Duration of pharmacologic treatment for neonatal abstinence syndrome up to 70 days of age
Measure: Median (Standard Deviation); unit: days
Arm/Group | Buprenorphine
Number analyzed (Participants) | 10
days | 30 (8.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected until infants were discharged from the hospital, an average of 30 days (range 11-42)
Description: definition of SAE matches that of clinicaltrials.gov
Arm/Group | Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=10)
seizure (Nervous system disorders) | 1 (1) — Seizure in setting of elevated Finnegan scores
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=10)
rash (Skin and subcutaneous tissue disorders) | 1 (1) — diffuse erythematous rash for 2 hours duration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03608696/Prot_000.pdf